CLINICAL TRIAL: NCT05394064
Title: A Phase 1/2 Randomized, Blinded, Dose-escalation Study to Evaluate the Safety and Efficacy of Intrathecal Administration of AAV9-ABCD1 Gene Therapy (SBT101) in Adult Patients With Adrenomyeloneuropathy
Brief Title: A Study to Evaluate Administration of SBT101 Gene Therapy in Adult Patients With Adrenomyeloneuropathy (AMN)
Acronym: PROPEL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The SBT101 program for AMN was terminated for business/strategic reasons, and there were no safety concerns
Sponsor: SwanBio Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBT101-CT101; 2021-004410-19 (EudraCT Number)
Record Dates: First submitted 2022-05-16; First posted 2022-05-27 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: AMN; AMN Gene Mutation; X-ALD
Keywords: AMN; X-ALD; Adrenoleukodystrophy; X-linked Adrenoleukodystrophy; Adrenomyeloneuropathy; Myeloneuropathy; Spastic paraplegia; Hereditary Spastic Paraplegia; HSP; ALD; ABCD1; ALDP; CALD; CCALD; Brain Diseases, Metabolic, Inborn; Brain Diseases, Metabolic; Hereditary Central Nervous System Demyelinating Diseases; Leukoencephalopathies; Demyelinating Diseases; Heredodegenerative Disorders, Nervous System; Metabolism, Inborn Errors; Peroxisomal Disorders; Metabolic Diseases; Adrenal Insufficiency; Gene Therapy; AAV9; Adeno-Associated Vector
MeSH Terms: conditions — Adrenoleukodystrophy; Paraplegia; Spastic Paraplegia, Hereditary; Brain Diseases, Metabolic, Inborn; Brain Diseases, Metabolic; Hereditary Central Nervous System Demyelinating Diseases; Leukoencephalopathies; Demyelinating Diseases; Heredodegenerative Disorders, Nervous System; Metabolism, Inborn Errors; Peroxisomal Disorders; Metabolic Diseases; Adrenal Insufficiency

STUDY DESIGN:
Intervention Model Description: 3 Cohorts, each with active treatment and 1 with imitation procedure
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Maintain masking to all but those are perform the actual procedure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): Patients treated with SBT101
  Interventions: Genetic: SBT101
- Imitation Procedure (Sham Comparator): Procedure that mimics treatment with SBT101, but does not infuse anything into the spinal cord
  Interventions: Procedure: Imitation Procedure

INTERVENTIONS:
Genetic: SBT101 — SBT101 Treatment
  Arms: Active Treatment
Procedure: Imitation Procedure — Procedure that mimics SBT101 infusion, but contains no drug administered
  Other Names: Sham Procedure
  Arms: Imitation Procedure

SUMMARY:
This is a Phase 1/2 randomized, blinded, dose-escalation study to evaluate the safety and efficacy of intrathecal (IT) administration of SBT101, a recombinant adeno-associated virus serotype 9 (AAV9) containing a functional copy of the human adenosine triphosphate (ATP)-binding cassette transporter subfamily D member 1 (ABCD1; hABCD1) gene, in adult patients with adrenomyeloneuropathy (AMN) aged 18-65 years.

Patients will receive a single dose of SBT101 via IT route (or an imitation procedure) and will be followed for safety and efficacy for 2 years. Patients receiving SBT101 will be followed for an additional 3 years (5 total) for Safety. Patients receiving an imitation procedure will be offered the opportunity to receive SBT101 after 2 years, as data indicate.

DETAILED DESCRIPTION:
The study consists of two parts after infusion of SBT101:

Part 1: A blinded 24-month core study period to evaluate the safety and potential impact of SBT101 on disease progression. Part 1 will consist of 2 phases:

Phase 1: Dose-Escalation Phase: Two (2) doses of SBT101 (Dose level 1 cohort and Dose Level 2 cohort) will be evaluated to establish the maximum tolerated dose (MTD).

Phase 2: Dose-Expansion Phase: Additional patients will be enrolled to receive SBT101 at the MTD

Part 2: An unblinded 3-year long-term safety follow-up period with annual follow-up visits to evaluate the safety of SBT101 and disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with X-linked adrenoleukodystrophy (ALD), including proven mutation in the ABCD1 gene through confirmatory genetic testing, and supported by elevated circulating VLCFA levels.
2. Clinical evidence of spinal cord involvement but still able to ambulate independently

Exclusion Criteria:

1. Evidence of or past diagnosis of inflammatory cerebral disease.
2. 15 years or more have elapsed since the initial onset of myeloneuropathy manifestations such as walking or running difficulties, bladder dysfunction, increased muscular tone, spasticity, weakness, balance problems, etc.
3. Contraindications for MRI procedure and/or contrast materials.
4. Contraindication to steroids, sirolimus, tacrolimus, and/or anesthetic medications.
5. Unstable adrenal function (e.g., untreated or inappropriately treated adrenal insufficiency).
6. History of diabetes or abnormal fasting plasma glucose (≥126 mg/dL) or hemoglobin A1C ≥6.5%.
7. Patients who have received a gene therapy.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on genetic gender
Enrollment: 8 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events to SBT101 | 2 years
  Safety and tolerability of SBT101 administration

SECONDARY OUTCOMES:
Disease progression | 2 years
  Characterize disease progression in adults diagnosed with AMN through serial clinical assessments of walking ability measured by 6-Minute Walk Test

OTHER OUTCOMES:
Change in Quality of Life | 2 years
  Characterize the change in multiple quality of life parameters over time using questionnaires including the Multiple Sclerosis Quality of Life-54 (MS-QOL)

CONTACTS AND LOCATIONS:
Locations (2):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States
- Amsterdam UMC, Amsterdam, Netherlands